CLINICAL TRIAL: NCT01548430
Title: A Double-blind, Randomized, Placebo-controlled, Phase 1 Study of 2 Escalating, Single Subcutaneous Doses to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of TTP4000 in Subjects With Alzheimer's Disease With Mild Cognitive Impairment
Brief Title: A Safety Study of TTP4000 in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: TTP4000-101
Record Dates: First submitted 2012-02-28; First posted 2012-03-08 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TTP4000 1.0 mg/kg (Experimental): Administered subcutaneously
  Interventions: Drug: TTP4000
- TTP4000 3.0 mg/kg (Experimental): Administered subcutaneously
  Interventions: Drug: TTP4000
- Placebo (Placebo Comparator): Administered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTP4000
  Arms: TTP4000 1.0 mg/kg; TTP4000 3.0 mg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to examine the safety, tolerability, immunogenicity and pharmacokinetics of TTP4000 in subjects with Alzheimer's disease with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 50 years of age.
* Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
* Weight ≥ 50 kg.
* Alzheimer's disease according to the DSM-IV-TR criteria and a score between 20 and 26 on the Mini Mental State Exam.
* Subject must have a medical history for at least 6 months prior to Screening (confirmed by medical records) of a diagnosis of mild Alzheimer's disease.

Exclusion Criteria:

* Current evidence or history within the last 3 years of a neurological or psychiatric illness that could contribute to dementia, including, but not limited to: epilepsy, focal brain lesion, Parkinson's disease, seizure disorder, or head injury with loss of consciousness; DSM-IV-TR criteria for any major psychiatric disorder, including psychosis, major depression, and bipolar disorder.
* Participation and dosing in another clinical trial, involving any marketed or investigational drug, within 30 days before Screening Visit.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of participant with adverse events | Day 0 to Day 84

SECONDARY OUTCOMES:
Evaluation of participant plasma TTP4000 concentrations | Day 0 to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hernandez, Ph.D., Study Director — TransTech Pharma, Inc.
Locations (3):
- United States (3):
  - Miami, Florida
  - Durham, North Carolina
  - High Point, North Carolina